CLINICAL TRIAL: NCT02837575
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Trial to Evaluate the Safety and Efficacy of Herpes Simplex Virus, Type 2 (HSV-2) Therapeutic DNA Vaccine in Adults With Symptomatic Genital HSV-2 Infection
Brief Title: Safety and Efficacy Study of Herpes Simplex Virus Type 2 (HSV-2) Therapeutic DNA Vaccine
Acronym: HSV-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSV2-201
Record Dates: First submitted 2016-07-13; First posted 2016-07-19 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Herpes Genitalis
Keywords: HSV-2; Genital Herpes; Herpes; Herpes Simplex Virus, Type 2
MeSH Terms: conditions — Herpes Genitalis; Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VCL-HB01, 1-mL dose (Experimental): VCL-HB01, 1-mL dose by intramuscular injection once every 28 days for 4 doses
  Interventions: Biological: VCL-HB01
- Phosphate-buffered saline, 1-mL dose (Placebo Comparator): PBS, 1-mL dose by intramuscular injection once every 28 days for 4 doses
  Interventions: Other: Phosphate-buffered saline

INTERVENTIONS:
Biological: VCL-HB01 — Investigational Product
  Arms: VCL-HB01, 1-mL dose
Other: Phosphate-buffered saline — Placebo
  Other Names: PBS
  Arms: Phosphate-buffered saline, 1-mL dose

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of a therapeutic DNA vaccine in adults with symptomatic herpes simplex virus type 2 (i.e., genital herpes).

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of 4 doses of VCL-HB01, a therapeutic HSV plasmid DNA vaccine formulated with Vaxfectin® in HSV-2-seropositive adults with a reported history of symptomatic genital herpes for at least one year.

ELIGIBILITY:
Inclusion Criteria:

* HSV-2 seropositive
* A minimum of 1 year of reported history of genital herpes with recurrences.

Exclusion Criteria:

* History of receiving an investigational HSV vaccine
* Chronic illness for which a subject's immune system is suspected to be impaired or altered, such as cancer, autoimmune conditions, or diabetes
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 261 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Lesion recurrences | Up to Day 450

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to Day 450
Time to first recurrence | Up to Day 450
Proportion of subjects recurrence-free | Up to Day 450

CONTACTS AND LOCATIONS:
Overall Officials: Mammen P Mammen, MD, FIDSA, Study Director — Vical
Locations (15):
- United States (15):
  - Alabama Vaccine Research Clinic at University of Alabama at Birmingham, Birmingham, Alabama
  - Medical Center for Clinical Research, San Diego, California
  - QPS Broward Research, Hollywood, Florida
  - QPS Miami Research Associates, South Miami, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - University of Illinois, Chicago, Illinois
  - Indiana University Infectious Disease Research, Indianapolis, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - University of North Carolina (UNC) Institute of Global Health and Infectious Diseases, Chapel Hill, North Carolina
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - University of Utah School of Medicine - Division of Infectious Diseases, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No